CLINICAL TRIAL: NCT04499560
Title: The Effects of a Nutrition Supplement on Health Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Collaborators: Young Living Essential Oils (Unknown)
Responsible Party: Principal Investigator, Jessie Hawkins, PhD, Research Director, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-7-1100
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Sleep; Stress; Health, Subjective; Inflammation; Cognitive Symptom
Keywords: immune health; prevention; phytonutrients; superfoods; antioxidant; essential oils
MeSH Terms: conditions — Inflammation; Neurobehavioral Manifestations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants consume 2 ounces of the supplement each morning for 60 days.
  Interventions: Dietary Supplement: Supplement Drink
- Control (No Intervention): Participants do not make any changes to their health related routines

INTERVENTIONS:
Dietary Supplement: Supplement Drink — Superfoods based nutritional supplement
  Arms: Intervention

SUMMARY:
The purpose of this study is to evaluate the health related benefits of a superfoods nutrition supplement on health related quality of life.

DETAILED DESCRIPTION:
After being informed about the study, participants will provide informed consent and be randomized to one of two groups: intervention or control. Those in the intervention group will consume two ounces of a superfoods drink each morning for 60 days. Outcomes will be assessed at baseline, on day 30 and on day 60.

ELIGIBILITY:
Inclusion Criteria:

* otherwise healthy
* adults living in the US
* is practicing adequate contraception or is abstaining from all activities which could result in pregnancy
* understands and agrees to comply with study procedures
* provides informed consent

Exclusion Criteria:

* smoker
* pregnant or may become pregnant
* currently breastfeeding
* currently taking antioxidant supplements
* underlying chronic health conditions
* COVID-19 diagnosis
* demonstrated inability to comply with study procedures
* history of allergy to citrus or berry fruits
* has participated in an interventional clinical study within 31 days prior to enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in sleep quality on Pittsburgh Sleep Quality Index (PSQI) on Day 60 | Baseline and day 60
  The PSQI is a validated, self reporting instrument assessing sleep. Possible scores range from 0 to 21 with higher scores indicating lower quality sleep. The instrument contains 19 items.
Change from baseline in general wellbeing on the Physical Health Questionnaire (PHQ) on Day 60 | Baseline and day 60
  The PHQ is a validated, self reporting instrument assessing general wellbeing through sleep, respiratory health, headache, and gastrointestinal symptoms. Possible scores on each item range from 1 to 7 with higher scores indicating greater frequency of symptoms. The instrument contains 14 items.
Change from baseline in cognitive wellness on the Self Report Measure of Cognitive Abilities (SRMCA) on Day 60 | Baseline and day 60
  The SRMCA is a validated, self reporting instrument assessing cognitive wellbeing. Possible scores range from 0 to 27 with higher scores indicating greater cognitive wellbeing. The instrument contains 44 items.
Number of days with any cold symptoms as defined by the Jackson Symptom Score on day 60. | Day 60
  The Jackson Symptom Score is a validated, self reporting instrument which contains 8 cold and flu symptoms. Scores range from 0 (no symptoms) to 8 (every one of the listed symptoms.)
Change from baseline in stress on the Perceived Stress Scale (PSS) on Day 60 | Baseline and Day 60
  The PSS is a validated, self reporting instrument assessing perceived stress. Possible scores range from 0 to 40 with higher scores indicating higher stress levels. The instrument contains ten items.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Hawkins, PhD, Principal Investigator — Nutraceuticals Research Institute
Locations (1):
- Franklin School of Integrative Health Sciences, Franklin, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No